CLINICAL TRIAL: NCT03672487
Title: Short-course Benznidazole Treatment to Reduce Trypanosoma Cruzi Parasitic Load in Women of Reproductive Age: A Non-inferiority Randomized Controlled Trial
Brief Title: Short-course Benznidazole Treatment to Reduce Trypanosoma Cruzi Parasitic Load in Women of Reproductive Age
Acronym: BETTY
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Tulane University School of Public Health and Tropical Medicine (Other)
Collaborators: Institute for Clinical Effectiveness and Health Policy (Other); University of California, San Diego (Other)
Responsible Party: Sponsor
Organization: Tulane University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R01HD095857 (NIH)
Record Dates: First submitted 2018-09-06; First posted 2018-09-14 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-04

CONDITIONS: Chagas Disease
Keywords: Congenital Transmission; Trypanosoma cruzi; Benznidazole
MeSH Terms: conditions — Chagas Disease | interventions — benzonidazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Placebo
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 60/300mg (Active Comparator): The investigators will use a preparation of benznidazole (BZN) that is commercially available in Argentina: Abarax® 100mg and 50mg tablets from ELEA laboratories (Buenos Aires, Argentina). The investigators will purchase the drug at full cost.
  Interventions: The standard 60d course will be 300 mg per day, which is similar to the dose used in the second phase of the BENEFIT trial. The drug will be administered orally in two doses per day: the standard course will be one 100mg and one 50mg tablet in the morning and in the evening for 60 days.
  Interventions: Drug: Benznidazole
- 30/150mg (Experimental): The investigators will use a preparation of benznidazole (BZN) that is commercially available in Argentina: Abarax® 100mg and 50mg tablets from ELEA laboratories (Buenos Aires, Argentina). ELEA laboratories will prepare the placebo oral tablets, which will be identical to the drug tablets in aspect and taste. The investigators will purchase the drug and placebo at full cost.
  Interventions: The BZN short course low dose scheme will be 150 mg per day for 30 days. The drug will be administered orally in two doses per day: the short course treatment will start with the active drug and then placebo oral tablet; one 100 mg tablet and one placebo tablet in the morning and one 50 mg tablet and one placebo tablet in the evening for the first 30 days. The last 30 days will be two placebo tablets in the morning and the evening.
  Interventions: Drug: Benznidazole; Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Benznidazole — Benznidazole tablet
  Other Names: Abarax
Drug: Placebo Oral Tablet — Sugar pill manufactured to mimic Benznidazole
  Other Names: Placebo (for Benznidazole)
  Arms: 30/150mg

SUMMARY:
The investigators are proposing to perform a double-blinded, non-inferiority randomized controlled trial comparing a short 30-day treatment with BZN 150mg/day (30d/150mg) vs. a 60-day treatment with BZN 300 mg/day (60d/300mg). The investigators will recruit not previously treated T. cruzi seropositive women with a live birth during the postpartum period in Argentina, randomize them at six months postpartum, and follow them up with the following specific aims:

Specific Aim 1: To measure the effect of BZN 30d/150mg compared to 60d/300mg preconceptional treatment on parasitic load measured by the frequency of positive PCR (primary outcome) and by real-time quantitative PCR (qPCR), immediately (Specific Aim 1a) and 10 months (Specific Aim 1b) after treatment.

Hypothesis 1a: The frequency of positive PCR and the parasitic load measured by qPCR immediately after BZN 30d/150mg will be non-inferior (Non Inferiority [NI] margin for PCR: 10% absolute difference) to BZN 60d/300mg.

Hypothesis 1b: The frequency of positive PCR and the parasitic load measured by qPCR 10 months after BZN 30d/150mg will be non-inferior (NI margin for PCR: 9% absolute difference) to BZN 60d/300mg.

Specific Aim 2: To measure the frequency of serious adverse events leading to treatment interruption of BZN 30d/150mg compared to 60d/300mg.

Hypothesis 2: The frequency of serious adverse events leading to treatment interruption will be 50% lower with BZN 30d/150mg than with BZN 60d/300mg.

A 24-month recruitment period is planned in four hospitals with 23,436 deliveries in 2015 and frequencies of T. cruzi seropositive women varying from 1.5% to 4.8%. The investigators are planning to enroll 600 T. cruzi seropositive women.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent from the mother.
* T. cruzi seropositivity confirmed by at least two positive tests.
* Live birth.

Exclusion Criteria:

* Women residing outside of the provinces of Chaco, Santiago del Estero, or Tucumán.
* Previous trypanocide treatment (BZN or nifurtimox).
* Female sterilization; no intention to use modern contraception methods during treatment.
* Positive pregnancy test.
* History of severe alcohol abuse within two years; renal insufficiency.

Min Age: 13 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Women of childbearing age
Enrollment: 273 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Frequency of positive PCR and the parasitic load measured by qPCR immediately after BZN 30d/150mg | 30 days for the 30d course arm, and 60 days for the 60d course arm
  The frequency of positive PCR and the parasitic load measured by qPCR immediately after BZN 30d/150mg will be non-inferior (Non Inferiority [NI] margin for PCR: 10% absolute difference) to BZN 60d/300mg.
The frequency of positive PCR and the parasitic load measured by qPCR 10 months after BZN 30d/150mg | 10 months from the end of the 60d treatment
  The frequency of positive PCR and the parasitic load measured by qPCR immediately after BZN 30d/150mg will be non-inferior (Non Inferiority [NI] margin for PCR: 10% absolute difference) to BZN 60d/300mg.

SECONDARY OUTCOMES:
The frequency of serious adverse events leading to treatment interruption of BZN 30d/150mg compared to 60d/300mg immediately after BZN 30d/150mg | 60 days after treatment initiation
  The frequency of serious adverse events leading to treatment interruption will be 50% lower with BZN 30d/150mg than with BZN 60d/300mg.

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Buekens, MD, PhD, Principal Investigator — Tulane University
Locations (3):
- United States (2):
  - University of California at San Diego, San Diego, California
  - Tulane School of Public Health and Tropical Medicine, New Orleans, Louisiana
- Institute for Clinical Effectiveness and Health Policy, Buenos Aires, Argentina

REFERENCES:
- [Derived] Cafferata ML, Toscani MA, Althabe F, Belizan JM, Bergel E, Berrueta M, Capparelli EV, Ciganda A, Danesi E, Dumonteil E, Gibbons L, Gulayin PE, Herrera C, Momper JD, Rossi S, Shaffer JG, Schijman AG, Sosa-Estani S, Stella CB, Klein K, Buekens P. Short-course Benznidazole treatment to reduce Trypanosoma cruzi parasitic load in women of reproductive age (BETTY): a non-inferiority randomized controlled trial study protocol. Reprod Health. 2020 Aug 24;17(1):128. doi: 10.1186/s12978-020-00972-1. PMID 32831069

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-20): https://cdn.clinicaltrials.gov/large-docs/87/NCT03672487/Prot_SAP_000.pdf